CLINICAL TRIAL: NCT06858670
Title: Effectiveness of Auxiliary Segmental Lingual Appliances in Leveling the Curve of Wilson at Second Molars
Acronym: EASLALCW
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hanoi Medical University (Other)
Responsible Party: Principal Investigator, Nguyen Ngoc Hoa, Principal Investigator, Hanoi Medical University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 240304
Record Dates: First submitted 2025-02-24; First posted 2025-03-05 (Actual); Last update posted 2025-03-05 (Actual); Status verified 2025-02

CONDITIONS: Malocclusion; Malocclusion; Displaced or Missing Teeth; Malocclusions; Orthodontic Treatment
Keywords: Auxiliary Segmental Lingual Appliances; Curve of Wilson; Second Molars; Labial Fixed Orthodontic Treatment; Split-Mouth Design; Digital Impressions; Malocclusion; Dental Occlusion; Orthodontic Treatment Outcomes
MeSH Terms: conditions — Malocclusion; Anodontia; Bites and Stings

STUDY DESIGN:
Masking Description: There will be no masking in this study. Both the patient and the outcome assessor will know which side will receive the intervention (auxiliary segmental lingual appliances).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Auxiliary Segmental Lingual Appliances Intervention in One Side (Experimental): In this arm, patients will receive the intervention of auxiliary segmental lingual appliances on one side of the mouth. The intervention aims to level the Curve of Wilson by adjusting the lingual inclination and leveling the lingual cusps of the mandibular second molar.
  Interventions: Procedure: Auxiliary Segmental Lingual Appliances
- Control in Another Side (No Intervention): In this arm, patients will not receive the intervention of auxiliary segmental lingual appliances on another side of the mouth.

INTERVENTIONS:
Procedure: Auxiliary Segmental Lingual Appliances — This intervention involves the use of auxiliary segmental lingual appliances specifically designed to level the Curve of Wilson at the second molars in patients undergoing labial fixed orthodontic treatment. The primary goal is to adjust the lingual inclination of the mandibular second molar, thereby achieving a more balanced and functional occlusal plane.
  Arms: Auxiliary Segmental Lingual Appliances Intervention in One Side

SUMMARY:
This study aims to evaluate the effectiveness of auxiliary segmental lingual appliances in leveling the Curve of Wilson at the second molars in patients undergoing labial fixed orthodontic treatment. Patients exhibiting an excessive (deep) Curve of Wilson at the second molar bilaterally (meaning lingually inclined mandibular second molar) will be recruited.. Using a split-mouth design, one side will receive the intervention (auxiliary segmental lingual appliances), while the other side will serve as the control. The variables measured include the Curve of Wilson at the second and first molars, and the distance from the mesiolingual and distolingual cusps of the second molar to the occlusal plane of the first molar. Measurements will be taken on digital impressions at baseline (T0), after leveling with a stainless steel labial archwire (T1), and three months after applying the auxiliary segmental lingual appliances. The effectiveness will be assessed by comparing the two groups.

DETAILED DESCRIPTION:
This study focuses on evaluating the effectiveness of auxiliary segmental lingual appliances in leveling the Curve of Wilson at the second molars in patients undergoing labial fixed orthodontic treatment. The study will recruit patients who exhibit an excessive (deep) Curve of Wilson at the second molar bilaterally (meaning lingually inclined mandibular second molar). A split-mouth design will be employed, where one side of the mouth will receive the intervention (auxiliary segmental lingual appliances), and the other side will serve as the control.

The primary variables measured include the Curve of Wilson at the second and first molars, and the distance from the mesiolingual and distolingual cusps of the second molar to the occlusal plane of the first molar. These measurements will be taken using digital impressions at three different time points: baseline (T0), after leveling with a stainless steel labial archwire (T1), and three months after the application of the auxiliary segmental lingual appliances.

The study aims to compare the effectiveness of the auxiliary segmental lingual appliances by analyzing the differences between the intervention and control sides. This comparison will help determine the impact of the appliances on achieving a more balanced and functional occlusal plane, potentially improving orthodontic treatment outcomes for patients with malocclusion issues.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing labial fixed orthodontic treatment.
* Patients exhibiting an excessive (deep) Curve of Wilson at the second molar bilaterally (meaning lingually inclined mandibular second molar).
* Patients willing to participate and provide informed consent.

Exclusion Criteria:

* Patients with limited mouth opening and gagging reflex preventing placement of auxiliary segmental lingual appliances.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-03-01 (Estimated); Primary Completion 2029-03-01 (Estimated); Study Completion 2029-03-01 (Estimated)

PRIMARY OUTCOMES:
Curve of Wilson at Second Molar | Baseline, 6 months, 9 months.
  This measure evaluates the angle between the occlusal plane of the second molar and the mandibular arch occlusal plane. Measurements will be taken using digital impressions.
Distance from Mesiolingual Cusp of Second Molar to Occlusal Plane of First Molar | Baseline, 6 months, 9 months.
  This measure evaluates the distance from the mesiolingual cusp of the second molar to the occlusal plane of the first molar. Measurements will be taken using digital impressions.
Distance from Distolingual Cusp of Second Molar to Occlusal Plane of First Molar | Baseline, 6 months, 9 months.
  Description: This measure evaluates the distance from the distoolingual cusp of the second molar to the occlusal plane of the first molar. Measurements will be taken using digital impressions.

SECONDARY OUTCOMES:
Curve of Wilson at First Molar | Baseline, 6 months, 9 months.
  Description: This measure evaluates the angle between the occlusal plane of the second molar and the mandibular arch occlusal plane. Measurements will be taken using digital impressions.

CONTACTS AND LOCATIONS:
Locations (1):
- Phenikaa University, Hanoi, Vietnam

IPD SHARING:
Plan to Share IPD: No